CLINICAL TRIAL: NCT05330286
Title: Randomized, Single-dose, Open-label, Two-part, Two-period, Cross-over Study to Compare the Pharmacokinetics, Safety and Tolerability of the Pediatric With an Adult Formulation of Branaplam and to Investigate the Adult Formulation in Fed and Fasted State in Healthy Participants
Brief Title: Study to Compare the Pharmacokinetics, Safety and Tolerability of the Pediatric and Adult Branaplam Formulation in Healthy Adults and the Effect of Food on the Latter.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The compound is no longer suitable for further clinical development due to a safety finding in a later phase program.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLMI070A02104
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Healthy Volunteers
Keywords: healthy; healthy participants; adult; Relative bioavailability study; branaplam; LMI070

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pediatric Formulation (Experimental): Part 1 - healthy participants receiving pediatric formulation
  Interventions: Drug: LMI070
- Adult Formulation (Experimental): Part 1 - healthy participants receiving adult formulation
  Interventions: Drug: LMI070
- Adult formulation fasted state (Experimental): Part 2- healthy participants receiving adult formulation in fasted conditions
  Interventions: Drug: LMI070
- Adult formulation Fed state (Experimental): Part 2- Part 2- healthy participants receiving adult formulation in fed conditions
  Interventions: Drug: LMI070

INTERVENTIONS:
Drug: LMI070 — oral solution
  Arms: Pediatric Formulation
Drug: LMI070 — Oral solution
  Arms: Adult Formulation
Drug: LMI070 — Oral solution given in fasted state
  Arms: Adult formulation fasted state
Drug: LMI070 — Oral solution given in fed state
  Arms: Adult formulation Fed state

SUMMARY:
This is a Phase 1 study designed to assess the relative bioavailability (BA), safety and tolerability and PK of the pediatric and adult formulations of branaplam.

DETAILED DESCRIPTION:
This study is to compare the pharmacokinetics, safety and tolerability of the pediatric and adult branaplam formulation in healthy adults. The study will also clarify if dosing with food can affect the PK of the adult formulation in order to guide recommendations on dosing relative to meals in subsequent studies. It is two-part, two-period, cross-over study in healthy participants which means that participants will receive both doses and take the treatment with and without food. The total study duration for each participant is expected to be up to approximately 88 days, including the Screening period and safety FU call.

Participants will be required to be stay at the site overnight for 6 days during each period to receive dose and have multiple blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and non-childbearing potential female participants, 18 to 60 years of age inclusive, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening and baseline 1 (laboratory parameters are listed in Table 8-4.
* Participants must weigh at least 50 kg at screening to participate in the study, and must have a body mass index within the range of 18.0 to 30.0 kg/m2 as measured at screening. Body mass index = Body weight (kg) / [Height (m)]2.
* At screening and baseline vital signs (systolic blood pressure, diastolic blood pressure and pulse rate) will be assessed in the supine position and again in the standing position (after at least 3 minutes in each position). Oral body temperature will also be taken with the other supine vital sign assessments. Supine vital signs must be within the following ranges at screening and baseline 1:

  * oral body temperature 35.0-37.5 °C (inclusive)
  * systolic blood pressure, 90-139 mmHg (inclusive)
  * diastolic blood pressure, 50-89 mmHg (inclusive)
  * pulse rate, 40-90 bpm (inclusive) Participants should be excluded if their standing vital signs (relative to supine) show findings which, in the opinion of the Investigator, are associated with clinical manifestation of postural hypotension (i.e. absence of any other cause). An Investigator should carefully consider enrolling participants with either a > 20 mmHg decrease in systolic blood pressure or a > 10 mmHg decrease in diastolic blood pressure accompanied by a > 20 bpm increase in pulse rate.

Exclusion Criteria:

* Participants who have received any investigational medicinal product in a clinical research study within the 90 days or 5 half-lives, whichever is longer, prior to Period 1 Day 1.
* Participants who have previously been administered investigational medicinal product in this study. Participants who have taken part in Part 1 are not permitted to take part in Part 2.
* Significant illness, which has not resolved within two (2) weeks prior to initial dosing.
* Men planning to father children in the near future (next 6 months).
* Male participant who reports to have a pregnant or nursing (lactating) partner.
* Sexually active males unwilling to adhere to the contraception requirements of the study as detailed below:

  * A condom is required for all sexually active male participants to prevent them from fathering a child AND to prevent delivery of the investigational drug via seminal fluid to their partner.
  * Males with partners of childbearing potential must use a condom during intercourse while taking investigational drug and for 118 days after stopping investigational drug (duration to cover one spermatogenesis cycle plus 5 half-lives).
  * Additionally, male participants with female partners of childbearing potential should also use another highly effective method of contraception. Highly effective contraception methods include:

Partner's bilateral tubal occlusion Male participant sterilization (vasectomy; at least 6 months prior to screening).

Partner's use of oral (estrogen and progesterone; or progesterone only that inhibits ovulation), injected, or implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system, or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months.

* Total abstinence (when this is in line with the preferred and usual lifestyle of the participant). Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Males with partners of non-childbearing potential must use a condom during intercourse while taking investigational drug and for 28 days after stopping investigational drug (duration to cover 5 half lives).
* In addition, male participants should not donate sperm for 118 days after stopping investigational drug.

  * Women of childbearing potential who report to be pregnant or nursing (lactating). Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant. Women are considered not of child-bearing potential if they are post-menopausal or have had surgical bilateral salpingectomy or bilateral oophorectomy (with or without hysterectomy) or total hysterectomy at least six weeks before screening. Women are considered post menopausal if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) and serum follicle stimulating hormone concentration of ≥40 IU/L. Follicle stimulating hormone and luteinizing hormone testing is required of any female participant, regardless of reported reproductive/menopausal status at screening. Refer to Section 8.4.3 Pregnancy and Assessments of Fertility.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Part 1: Plasma Cmax | Day 1, 2, 3, 4, 5, 8, 11 and 15
  Assess relative bioavailability of adult vs pediatric formulation of branaplam under fasting conditions
Part 1: Plasma AUClast | Day 1, 2, 3, 4, 5, 8, 11 and 15 in each period
  Assess relative bioavailability of adult vs pediatric formulation of branaplam under fasting conditions
Part 1: Plasma AUCinf | Day 1, 2, 3, 4, 5, 8, 11 and 15 in each period
  Assess relative bioavailability of adult vs pediatric formulation of branaplam under fasting conditions
Part 2:Plasma Cmax | Day 1, 2, 3, 4, 5, 8, 11 and 15 in each period
  Investigate food effect on the pharmacokinetics of the adult formulation of branaplam
Part 2: Plasma AUClast | Day1, 2, 3, 4, 5, 8, 11 and 15 in each period
  Investigate food effect on the pharmacokinetics of the adult formulation of branaplam
Part 2: Plasma AUCinf | Day 1, 2, 3, 4, 5, 8, 11 and 15 in each period
  Investigate food effect on the pharmacokinetics of the adult formulation of branaplam

SECONDARY OUTCOMES:
Number of Adverse events and Serious adverse events | Day 1 up to 30 days after last drug administration
  Any clinically significant events from other safety assessments will be recorded as adverse events as evaluated by investigator.
Parts 1 & 2: Plasma Cmax | Day 1, 2, 3, 4, 5, 8, 11 and 15 in each period
  Assess the Pharmacokinetic profile of branaplam and its metabolite UFB112
Parts 1 & 2: Plasma AUClast | Day 1, 2, 3, 4, 5, 8, 11 and 15 in each period
  Assess the Pharmacokinetic profile of branaplam and its metabolite UFB112
Parts 1 &2: Plasma AUCinf | Day 1, 2, 3, 4, 5, 8, 11 and 15 in each period
  Assess the Pharmacokinetic profile of branaplam and its metabolite UFB112
Parts 1 & 2: Plasma Tmax | Day 1, 2, 3, 4, 5, 8, 11 and 15 in each period
  Assess the Pharmacokinetic profile of branaplam and its metabolite UFB112
Parts 1 & 2: T1/2 | Day 1, 2, 3, 4, 5, 8, 11 and 15 in each period
  Assess the Pharmacokinetic profile of branaplam and its metabolite UFB112
Parts 1 & 2: Plasma Vz/F | Day 1, 2, 3, 4, 5, 8, 11 and 15 in each period
  Assess the Pharmacokinetic profile of branaplam and its metabolite UFB112
Parts 1 & 2: Plasma CL/F | Day 1, 2, 3, 4, 5, 8, 11 and 15 in each period
  Assess the Pharmacokinetic profile of branaplam and its metabolite UFB112

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Mere Way, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.